CLINICAL TRIAL: NCT02164500
Title: A Phase II, Open-label, Prospective, Non-randomized, Multicenter Clinical Trial With the JAK-inhibitor Ruxolitinib in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: JAK-inhibition in Recurrent Classical Hodgkin Lymphoma
Acronym: JeRiCHO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Bastian von Tresckow, Dr., University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JeRiCHO
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Recurrent Classical Hodgkin Lymphoma
MeSH Terms: interventions — ruxolitinib

ARMS (1):
- Ruxolitinib (Experimental)
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib

SUMMARY:
The Purpose of this trial is:

* to determine the overall response rate (ORR, complete response [CR] + partial response [PR]) in patients with relapsed or refractory HL
* to determine the safety profile of ruxolitinib in patients with relapsed or refractory HL

ELIGIBILITY:
Inclusion Criteria:

* relapsed or refractory HL
* ECOG <= 2,
* no major organ dysfunction
* written informed consent

Exclusion Criteria:

* history of another primary malignancy ≤ 2 years
* female patients who are pregnant or breast feeding
* patients with a known history of HIV seropositivity
* chronic active hepatitis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
overall response rate | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Dept. of Medicine, Cologne University Hospital, Cologne, Germany

REFERENCES:
- See also: Homepage GHSG — http://www.ghsg.org